CLINICAL TRIAL: NCT06837493
Title: Investigation of the Effects of Different Rehabilitation Approaches on Cognitive Functions, Dual Task Performance, and Manual Dexterity in Older Adults With Mild Cognitive Impairment
Brief Title: Investigation of Different Rehabilitation Approaches in Older Adults With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Kevser Gürsan, Principal Investigator, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 210023
Record Dates: First submitted 2025-02-05; First posted 2025-02-20 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment (MCI); Geriatric
Keywords: Mild cognitive impairment; hand exercises; cognitive training; hand functions; cognitive functions
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hand exercise group (HEG) (Experimental): The first experimental group received resistance-based hand exercises and functional task-oriented hand exercise group (HEG)
  Interventions: Other: Resistance based hand exercises and functional task-oriented hand exercise
- Cognitive training group (CTG) (Experimental): The second experimental group received cognitive training group (CTG)
  Interventions: Other: Cognitive training
- Control group (CG) (No Intervention): The control group (CG) did not receive any training and continued with their daily routines

INTERVENTIONS:
Other: Resistance based hand exercises and functional task-oriented hand exercise — The interventions for HEG were administered by a physiotherapist over a period of eight weeks, with three sessions conducted each week.
  Arms: Hand exercise group (HEG)
Other: Cognitive training — The interventions for CTG were administered by a physiotherapist over a period of eight weeks, with three sessions conducted each week.
  Arms: Cognitive training group (CTG)

SUMMARY:
This randomized controlled trial aims to comparatively examine whether cognitive training and hand exercise training provided to older adults with mild cognitive impairment (MCI) have an impact on their cognitive functions, hand skills, grip strength, activities of daily living, dual task performance, and interactions. Based on the study's objectives, the following hypotheses were formulated:

* Hypothesis 1: Cognitive training has an effect on cognitive functions in older adults with MCI.
* Hypothesis 2: Cognitive training has an effect on dual-task performance in older adults with MCI.
* Hypothesis 3: Cognitive training has an effect on hand skills in older adults with MCI.
* Hypothesis 4: Resistance based hand exercises and functional task-oriented hand exercise training have an effect on cognitive functions in older adults with MCI.
* Hypothesis 5: Resistance based hand exercises and functional task-oriented hand exercise training have an effect on dual-task performance in older adults with MCI.
* Hypothesis 6: Resistance-based hand exercises and functional task-oriented hand exercise training have an effect on hand skills in older adults with MCI.

In this study, two different exercise interventions were applied to two experimental groups of individuals with mild cognitive impairment, while the control group did not receive any intervention. The first experimental group (Hand Exercise Group, HEG) and the second experimental group (Cognitive Training Group, CTG) underwent training administered by a physiotherapist three times per week for eight weeks.

To ensure assessor blinding, pre- and post-intervention assessments of the participants were conducted by an independent expert physiotherapist who was not involved in the study. The sociodemographic characteristics of the participants were collected using a data collection form. Cognitive functions were assessed with the Montreal Cognitive Assessment (MoCA); hand dominance was determined using the Edinburgh Handedness Inventory (EHI); hand dexterity was evaluated with the Nine-Hole Peg Test (NHPT); grip strength was measured using a hand dynamometer; motor-motor dual task performance (MMDTP) and motor-cognitive dual task performance (MCDTP) were assessed using a stopwatch; activities of daily living were evaluated with the Manual Ability Measurement-36, (MAM-36); and dual task interaction (DTI) was calculated using the following formula: DTI = (Single Task Performance - Dual Task Performance) / Single Task Performance × 100%.

DETAILED DESCRIPTION:
The number of individuals aged 65 and older is increasing worldwide, leading to a rise in the elderly population. As this demographic grows, the prevalence and diversity of health problems associated with aging are also increasing. The most common health issues in aging individuals include cognitive impairments, dementia, cardiovascular diseases, arthritis, type 2 diabetes mellitus (DM), and cancer.

The primary underlying causes of the frequent health problems in elderly individuals stem from negative changes in their physical, psychosocial, and cognitive conditions. Notably, structural, physiological, and functional declines in cognitive domains significantly impact the lives of elderly individuals. Cognitive function encompasses a broad range of processes and structures, including emotion, memory, reasoning, language, sensory processing, comprehension, analysis, interpretation, learning, and motor skills. Aging leads to structural deterioration, functional decline, dysfunction, and eventual loss of these cognitive abilities, contributing to various levels of cognitive impairment in elderly individuals. Depending on the severity and the affected cognitive domains, aging individuals may develop different neurological disorders. The most prevalent neurological conditions associated with aging include Mild Cognitive Impairment (MCI), Alzheimer's disease (AD), Parkinson's disease (PD), multiple system atrophy, Lewy body dementia, amyotrophic lateral sclerosis (ALS), progressive supranuclear palsy, and frontotemporal dementia.

Mild Cognitive Impairment is characterized by memory loss or other cognitive deficits that are not severe enough to interfere with daily activities but represent a transitional phase between normal cognitive function and early dementia. Other cognitive deficits include attention, sensory processing, language, visual-spatial perception, praxis, and motor skills. In elderly individuals with MCI, the type and severity of cognitive impairment vary depending on the affected structures within the central nervous system. Although these cognitive impairments manifest at different levels, most elderly individuals with MCI can still perform many daily activities independently.

Motor functions are defined as learned skills aimed at achieving specific goals, with hand motor skills involving a series of complex movements. Hand movement is directly linked to the motor and somatosensory homunculus through short U-shaped fibers that pass beneath the central sulcus. The distribution of these short U-shaped fibers follows the topographic organization of the primary motor and somatosensory cortex. Compared to other body regions, there are greater interconnections between finger regions, and the cortical areas allocated for tactile and proprioceptive information from the fingers are more extensive than those for other body parts.

The neuronal connections that maintain and support the functionality of fine and gross motor skills of the hand interact with the cortical areas of the brain. Therefore, any degenerative changes in these neuronal connections and cortical areas may influence individuals' cognitive and motor functions. The cortical areas of the brain govern high-level cognitive functions such as attention, thought, memory, perception, reasoning, awareness, coordination, language, comprehension, and speech. The relationship between cognitive functions and hand skills is still a topic of debate.

The relationship between cognitive functions and hand skills is explained through two primary mechanisms. The first mechanism suggests that cognitive and motor processes within the central nervous system share common neural pathways and are influenced by the same neural processes. In other words, the neural circuitry responsible for hand motor functions may be associated with cognitive performance. The second mechanism explaining the relationship between cognitive functions and hand skills involves the aging-related decline in the frontal lobe, particularly in the frontoparietal and frontostriatal areas, which are responsible for higher-level cognitive functions. These areas play a crucial role in motor control of the upper extremities and are actively engaged in fine and gross motor activities. Therefore, improving gross and fine motor performance of the upper extremities may enhance cognitive functions in elderly individuals by stimulating the frontal lobe.

Based on this perspective, our study aims to explore the relationship between cognitive functions and hand skills by implementing hand exercises and cognitive training in different groups of elderly individuals with MCI. The literature includes few studies investigating the connection between cognitive function and hand function. Therefore, this study seeks to examine the effects of different training interventions on cognitive functions, hand skills, grip strength, daily living activities, dual-task performance, and interaction in elderly individuals with MCI.

As part of the study, elderly individuals with MCI will undergo cognitive training and hand exercise programs. The hand exercise programs will include functional task-oriented and resistance-based hand exercises. No prior study in the literature has comprehensively examined the impact of such interventions on cognitive functions, hand skills, daily living activities, dual-task performance, and interaction in elderly individuals with MCI.

The primary objective of this study is to comparatively evaluate the effects of cognitive training and hand exercise programs on cognitive functions, hand skills, grip strength, daily living activities, dual-task performance, and interaction in elderly individuals with MCI.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years of age or older.
* Volunteering for the training.
* Scoring between 16-20 on the Montreal Cognitive Assessment.
* Being at least literate.

Exclusion Criteria:

* Having severe auditory and visual impairments.
* Having an unstable chronic condition (e.g., acute myocardial infarction, advanced respiratory distress requiring oxygen supplementation).
* Having Pulmonary Hypertension, dementia, hypertension , or brain damage.
* Having a history of major surgery within the last six months.
* Having upper extremity disorders (e.g., severe shoulder, elbow, wrist, finger, or bilateral elbow/wrist fractures, or advanced rheumatoid arthritis).

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Cognitive Functions | 8 weeks
  The Montreal Cognitive Assessment (MoCA) was used to assess the cognitive functions of the cases. The MoCA was administered through a face-to-face interview method, and the assessment took approximately 7 to 10 minutes to complete. The maximum possible score on the scale is 30 points. A score of 21 or higher is considered indicative of normal and healthy cognitive function, while scores between 16 and 20 indicate mild cognitive impairment, and a score of 15 or lower suggests dementia.
  The MoCA was chosen for this study due to its higher sensitivity in detecting cognitive impairment compared to other assessment tools.
Assessment of Hand Grip Strength | 8 weeks
  The hand grip strength of the participants was measured using a Takei hand dynamometer (T.K.K. 5101 model, Takei Scientific Instruments Co., Ltd, Tokyo, Japan). During the measurement, participants were seated in an upright position. Special attention was given to ensuring that the chair used had no armrests. The shoulder was positioned in adduction and neutral alignment, while the elbow and knee angles were adjusted to 90 degrees. The wrist was placed in a neutral position before the measurements were taken.
  Each participant performed three consecutive measurements using the Takei hand dynamometer, and the average of the three values was recorded as the final grip strength score. Measurements were conducted for both hands (right and left).
  The Takei hand dynamometer was selected as the assessment tool due to its validity and reliability in measuring hand grip strength and its easy
Assessment of Manual Dexterity | 8 weeks
  The Nine Hole Peg Test (NHPT) was administered to assess the participants' manual dexterity. The NHPT consists of a platform with nine holes and nine peg. The NHPT platform was positioned directly in front of the participants. During the test, the participants' body posture was carefully controlled: they were seated with their feet in contact with the floor, their backs supported by a chair, and their hips and knees at a 90° flexion position. Participants were informed that they could use their non-dominant hand to support the platform while performing the task.
  After explaining the rules of the NHPT, the participants were instructed to practice before starting the actual test. The task required the participants to insert the pegs into the holes as quickly as possible and then remove the pegs and place them into a box. Test results were recorded by timing the task using a stopwatch.

SECONDARY OUTCOMES:
Assessment of Dual Task Performance | 8 weeeks
  The Dual Task Performance (DTP) was assessed separately for both motor motor dual task performance (MMDTP) and motor cognitive dual task performance (MCDTP) for each hand (right and left) of the participants.
Assessment of Dual-Task Interaction (DTI) | 8 weeks
  Dual Task Interaction (DTI) is calculated by determining the difference between the single task performance time (time taken to perform the NHPT) and the dual task performance time (time taken to perform both the motor and cognitive tasks). The following formula was used to calculate the Motor Motor Dual Task Interaction (MMDTI) and Motor Cognitive Dual Task Interaction (MCDTI), and the times for each participant were recorded. The overall DTI evaluation for each participant was calculated using the following formulas:
  DTI = (Single Task Performance - Dual Task Performance) / Single Task Performance × 100.
  MMDTI = (Single Task Performance - MMDTP) / Single Task Performance × 100. MCDTI = (Single Task Performance - MCDTP) / Single Task Performance × 100.
Assessment of the Impact of Activities of Daily Living | 8 weeks
  Manual Ability Measurement-36, (MAM-36) was used to evaluate the impact of hand function on activities of daily living. MAM-36 is a self-reported assessment tool that evaluates functional limitations based on the participants' perceptions and responses.The scale focuses on functionality and incorporates participants' perceptions. The tasks in the MAM-36 represent various daily activities commonly performed in everyday life. The MAM-36 is comprised of clear and simple instructions, focusing on the functional capacity of a single hand.The Manual Ability Measure-36 (MAM-36) scoring system ranges from 0 to 100. Higher scores (closer to 100): Indicate better manual ability and minimal functional limitations in daily activities. Lower scores (closer to 0): Represent greater difficulties in performing daily tasks due to impaired hand function.

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Gursan, Dr., Principal Investigator — Uşak University
Locations (1):
- Elderly Care and Nursing Homes in Yozgat Province, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gursan K, Bayar K. Investigation of the effects of different rehabilitation approaches in elderly individuals with mild cognitive impairment. BMC Geriatr. 2026 Jan 10;26(1):185. doi: 10.1186/s12877-025-06946-x. PMID 41519716